CLINICAL TRIAL: NCT05576194
Title: Effect of Intraoperative Topical Application of a Taurolidine Solution on CIED Related Infections in the Clinical Setting - a Prospective Observational Study With a Restrospective Historical Control
Brief Title: Taurolidine Containing Antimicrobial CIED Wash to Prevent Infection
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Hendrik Bonnemeier (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Hendrik Bonnemeier, Coordinating principal investigator, University of Kiel
Organization: University of Kiel (Other)
Other Study IDs: 19059
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Implantable Electronic Device Infection
Keywords: cardiac implantable electronic device infection, taurolidine
MeSH Terms: interventions — taurolidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TauroPace irrigation group: every consecutive CIED placement, revision, extraction conducted with TauroPace
  Interventions: Device: TauroPace
- antiseptic irrigation group: every procedure conducted with adjunct antiseptic irrigation, which could be Taurolidine, TauroPace or Hydrogen Peroxide 3%
  Interventions: Device: TauroPace; Device: Hydrogen Peroxide; Drug: Taurolidine

INTERVENTIONS:
Device: TauroPace — All the hardware (leads, suture sleeves, pulse generator) is washed and the device pocket irrigated with an adjunct antimicrobial solution containing Taurolidine (TauroPace™, Tauropharm, Bavaria, Germany), during any invasive procedure (new implantation, pulse generator replacement, lead repositioning or insertion, system upgrade or downgrade, revision) involving a CIED system since January 2019
Device: Hydrogen Peroxide — All the hardware (leads, suture sleeves, pulse generator) was washed and the device pocket irrigated with an adjunct antimicrobial solution containing 3% hydrogen peroxide (H2O2) during any invasive procedure (new implantation, pulse generator replacement, lead repositioning or insertion, system upgrade or downgrade, revision) involving a CIED system at the authors' institute before 01/01/2020
  Groups: antiseptic irrigation group
Drug: Taurolidine — All the hardware (leads, suture sleeves, pulse generator) was washed and the device pocket irrigated with an adjunct antimicrobial solution containing taurolidine in a galenic formulation during any invasive procedure (new implantation, pulse generator replacement, lead repositioning or insertion, system upgrade or downgrade, revision) involving a CIED system at the authors' institute before 01/01/2019
  Groups: antiseptic irrigation group

SUMMARY:
From January 1st 2020, any CIED procedure conducted with adjunct TauroPace™ CIED and pocket irrigation is enrolled in a consecutive manner and followed up in one centre. Follow-up is prospectively.

Before that date any CIED procedure conducted with adjunct antispetic pocket and CIED irrigation is evaluated retrospectively to form a comparable group.

DETAILED DESCRIPTION:
All the hardware (leads, suture sleeves, pulse generator) is washed and the device pocket irrigated with an adjunct antimicrobial solution, which could be 3% hydrogen peroxide (H2O2), taurolidine in a galenic formulation or TauroPace™ (TP, Tauropharm, Bavaria, Germany), during any invasive procedure (new implantation, pulse generator replacement, lead repositioning or insertion, system upgrade or downgrade, revision) involving a CIED system at the authors' institute. Before 01/01/2020, the choice of antimicrobial solution was at the operator's discretion. These procedures were evaluated retrospectively. With change of policy on the first of January 2020, in every consecutive patient and procedure only TP is used. Patients were enrolled and followed consecutively in order of appearance. All CIED procedures performed at the author's institute between 01/01/2017 and 28/02/2022 are included for analysis. Patients who receive the galenic taurolidine formulation were excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

CIED procedure, signs PIC

Exclusion Criteria:

PIC not signed, minor

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The intervention group consists of every consecutive patient eligible for any CIED related surgical procedure in the centre of the investigation from January 2020 through February 2022 onwards.
Sampling Method: Non-Probability Sample
Enrollment: 1417 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
CIED infection | three months
  cardiac implantable electronic device infection

SECONDARY OUTCOMES:
all cause mortality | three months
  death of any cause during the observation
adverse events grade 3-5 | three months
  adverse events related to CIED, procedure or the atiseptic used
all cause mortality | 36 months
  death of any cause during all of the follow up period
adverse events grade 3-5 | 36 months
  adverse events related to CIED, procedure or the atiseptic used during all of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Borov, MD, Principal Investigator — Lakumed Landshut, CAU Kiel
Locations (1):
- Lakumed, Landshut, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borov, S., Baldauf, B., Lau, E.W. et al. Salvage of infected cardiac implantable electronic device with taurolidine-a case report. Cardiothorac Surg 30, 7 (2022). https://doi.org/10.1186/s43057-022-00068-5
- [Background] Giaccardi M, Baldauf B, Lau EW, Borov S, Bonnemeier H. Salvage of Cardiac Implantable Electronic Device Pocket Infection with Skin Erosion in Frail 92-Year-Old. J Cardiovasc Dev Dis. 2022 Mar 10;9(3):81. doi: 10.3390/jcdd9030081. PMID 35323629
- [Background] Weichsel J, Baldauf B, Bonnemeier H, Lau EW, Dittrich S, Cesnjevar R. Eradication of Ventricular Assist Device Driveline Infection in Paediatric Patients with Taurolidine. J Cardiovasc Dev Dis. 2022 Jan 10;9(1):18. doi: 10.3390/jcdd9010018. PMID 35050228
- [Derived] Borov S, Baldauf B, Henke J, Pavaci H, Perani A, Zrenner B, Dietl J, Mehilli J, Lau EW, Vonthein R, Bonnemeier H. Use of a taurolidine containing antimicrobial wash to reduce cardiac implantable electronic device infection. Europace. 2023 Oct 5;25(10):euad306. doi: 10.1093/europace/euad306. PMID 37831737